CLINICAL TRIAL: NCT05594420
Title: Bleeding and Needs for Blood Transfusion in Mitral Valve Replacement, Comparison Between Median Sternotomy and Minimally Invasive Approach.
Brief Title: Bleeding and Blood Transfusion in MVR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mustafa Loay Mohammed, Resident Doctor, Assiut University
Other Study IDs: Bleeding in MVR
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Mitral Valve Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MVR through Median sternotomy
  Interventions: Procedure: Mitral valve replacement
- MVR through Minimally invasive approach
  Interventions: Procedure: Mitral valve replacement

INTERVENTIONS:
Procedure: Mitral valve replacement — Mitral valve replacement through median sternotomy and minimally invasive approach

SUMMARY:
To identify the best approach for mitral valve replacement to decrease risk of bleeding and restrict blood transfusion and its complication.

DETAILED DESCRIPTION:
Mitral valve disease is the most common form of the valvular heart disorders including mitral regurgitation and mitral stenosis. Surgical treatment includes repair and replacement with different approaches as conventional median sternotomy or minimally invasive approaches.

Since minimally invasive mitral valve surgery (MMVS) was first described in the mid-to-late 1990s by pioneer surgeons Alain Carpentier and Randolph Chitwood, the techniques have evolved to include mini-thoracotomy, port-access thoracoscopic, partial sternotomy, and robotic. Right lateral mini-thoracotomy has become the standard approach for mitral valve surgery in many centers. These approaches may result in less surgical trauma, blood transfusions, and pain, thereby leading to a shorter hospital stay and faster return to daily activities. A reduction in postoperative hemorrhage and transfusion requirements have been suggested as a potential advantage of minimally invasive valve surgery. This benefit is important given the significant morbidity and mortality associated with transfusions and re-exploration for bleeding. Observational studies suggested that patients undergoing MMVS required fewer units of pRBCs transfused per patient and patients were at lower risk of transfusion. RCTs did not reach statistical significance. So, more studies were required to reach a definite conclusion.

Through this study our aim is to evaluate postoperative bleeding and needs for blood transfusion in conventional median sternotomy mitral valve replacement in comparison to minimally invasive approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mitral valve replacement through minimally invasive or median sternotomy at Assiut Cardiothoracic surgery department.

Exclusion Criteria:

* Patients refused to be enrolled in research. Emergency, redo procedures, active infectious endocarditis, and combined surgery (valve surgery and coronary artery bypass graft).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18-80 years old, males or females, undergoing mitral valve replacement through minimally invasive or median sternotomy at Assiut Cardiothoracic surgery department.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
bleeding | Baseline
  Amount of post operative bleeding per drains
Blood transfusion | Baseline
  Amount of blood products transfused

SECONDARY OUTCOMES:
Reexploration | Baseline
  Number of patients re-explored due to massive bleeding
Complications of blood transfusion | Baseline
  Complications of blood transfusion
ICU stay | Baseline
  Numbered of days patient stayed in ICU
Cost effectiveness | Baseline
  Financial aspect

REFERENCES:
- [Background] Nishimura RA, Vahanian A, Eleid MF, Mack MJ. Mitral valve disease--current management and future challenges. Lancet. 2016 Mar 26;387(10025):1324-34. doi: 10.1016/S0140-6736(16)00558-4. PMID 27025438
- [Background] Carpentier A, Loulmet D, Carpentier A, Le Bret E, Haugades B, Dassier P, Guibourt P. [Open heart operation under videosurgery and minithoracotomy. First case (mitral valvuloplasty) operated with success]. C R Acad Sci III. 1996 Mar;319(3):219-23. French. PMID 8761668
- [Background] Sundermann SH, Sromicki J, Rodriguez Cetina Biefer H, Seifert B, Holubec T, Falk V, Jacobs S. Mitral valve surgery: right lateral minithoracotomy or sternotomy? A systematic review and meta-analysis. J Thorac Cardiovasc Surg. 2014 Nov;148(5):1989-1995.e4. doi: 10.1016/j.jtcvs.2014.01.046. Epub 2014 Feb 5. PMID 24589199
- [Background] Al Otaibi A, Gupta S, Belley-Cote EP, Alsagheir A, Spence J, Parry D, Whitlock RP. Mini-thoracotomy vs. conventional sternotomy mitral valve surgery: a systematic review and meta-analysis. J Cardiovasc Surg (Torino). 2017 Jun;58(3):489-496. doi: 10.23736/S0021-9509.16.09603-8. Epub 2016 Sep 2. PMID 27588617
- [Background] Modi P, Hassan A, Chitwood WR Jr. Minimally invasive mitral valve surgery: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2008 Nov;34(5):943-52. doi: 10.1016/j.ejcts.2008.07.057. Epub 2008 Sep 30. PMID 18829343
- [Background] Eqbal AJ, Gupta S, Basha A, Qiu Y, Wu N, Rega F, Chu FV, Belley-Cote EP, Whitlock RP. Minimally invasive mitral valve surgery versus conventional sternotomy mitral valve surgery: A systematic review and meta-analysis of 119 studies. J Card Surg. 2022 May;37(5):1319-1327. doi: 10.1111/jocs.16314. Epub 2022 Feb 16. PMID 35170791